CLINICAL TRIAL: NCT00822081
Title: Comparison of the Fixed Combinations of Brimonidine/Timolol and Dorzolamide/Timolol in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bp Consulting, Inc (Network)
Collaborators: Allergan (Industry)
Responsible Party: Therapeutic Area Hand, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COM0501
Record Dates: First submitted 2009-01-12; First posted 2009-01-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Brimonidine Tartrate; Timolol; Brimonidine Tartrate, Timolol Maleate Drug Combination; dorzolamide; dorzolamide-timolol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): brimonidine/timolol. Fixed-combination monotherapy.
  Interventions: Drug: brimonidine tartrate 0.2%/timolol maleate 0.5% fixed combination
- 2 (Active Comparator): dorzolamide/timolol. Fixed-combination monotherapy.
  Interventions: Drug: dorzolamide hcl 2%/ timolol maleate 0.5% fixed combination
- 3 (Active Comparator): prostaglandin analogue+ brimonidine/timolol fixed combination.
  Interventions: Drug: brimonidine tartrate 0.2%/timolol maleate 0.5% fixed combination as adjunctive to current prostaglandin therapy.
- 4 (Active Comparator): prostaglandin analogue+dorzolamide/timolol fixed combination.
  Interventions: Drug: dorzolamide hcl 2%/timolol maleate 0.5% fixed combinatin as adjunctive to current prostaglandin therapy.

INTERVENTIONS:
Drug: brimonidine tartrate 0.2%/timolol maleate 0.5% fixed combination — 1 drop BID in each eye
  Other Names: Combigan.
  Arms: 1
Drug: dorzolamide hcl 2%/ timolol maleate 0.5% fixed combination — 1 drop BID in each eye
  Other Names: Cosopt.
  Arms: 2
Drug: brimonidine tartrate 0.2%/timolol maleate 0.5% fixed combination as adjunctive to current prostaglandin therapy. — 1 drop BID in each eye
  Other Names: Combigan.
  Arms: 3
Drug: dorzolamide hcl 2%/timolol maleate 0.5% fixed combinatin as adjunctive to current prostaglandin therapy. — 1 drop BID in each eye
  Other Names: Cosopt
  Arms: 4

SUMMARY:
This study compares the efficacy and tolerability/comfort of brimonidine/timolol and dorzolamide/timolol in patients with open-angle glaucoma or ocular hypertension. In an investigator masked randomization process, each subject is allocated to recieve either brimonidine/timolol or dorzolamide/timolol as fixed-combination monotherapy or as an adjuctive to a prostoglandin analogue for a period of 12 weeks. After screening, patient returns at baseline, Month 1, and Month 3 for ophthalmic evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 yrs.
* Female subjects of childbearing potential must have negative pregnancy test and provide contraception.
* Subjects must have confirmed diagnosis of primary open-angle glaucoma or ocular hypertension in both eyes.
* Subjects who are or have been insufficiently responsive to IOP reducing monotherapy and use of either study medication is deemed appropriate.
* Subjects able to complete questionnaires and provide informed consent.

Exclusion Criteria:

* Female subjects who are pregnant, planning to become pregnant during study period, breast feeding or not practicing a reliable method of birth control.
* Subjects wherein the study drugs are containdicated.
* Subjects who have had introcular surgery with 6 months (3 months for laser).
* Subjects with known side effects/ allergy or sensitivity to any component of study treatments.
* Subjects with any uncontrolled systemic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2005-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean IOP. | 12 weeks

SECONDARY OUTCOMES:
Patient tolerability/comfort measured by Likert scale. | Month 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Barrie, Ontario, Canada

REFERENCES:
- [Derived] Nixon DR, Yan DB, Chartrand JP, Piemontesi RL, Simonyi S, Hollander DA. Three-month, randomized, parallel-group comparison of brimonidine-timolol versus dorzolamide-timolol fixed-combination therapy. Curr Med Res Opin. 2009 Jul;25(7):1645-53. doi: 10.1185/03007990902994041. PMID 19476406